CLINICAL TRIAL: NCT01323257
Title: A Phase I, 2-panel, Open-label, Randomized, Crossover Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC435 and CYP3A Inhibitors, Erythromycin and Darunavir/Ritonavir (DRV/r)
Brief Title: TMC435-TiDP16-C115 - A Study in Healthy Volunteers Investigating the Pharmacokinetic Interaction Between TMC435 and Erythromycin and Between TMC435 and Darunavir/Ritonavir (DRV/r)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR018010; TMC435-TiDP16-C115
Record Dates: First submitted 2011-03-10; First posted 2011-03-25 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C115; TMC435-C115; TMC435; HCV; Hepatitis C; Hep C; healthy volunteers
MeSH Terms: conditions — Hepatitis C | interventions — Erythromycin; Ritonavir; Simeprevir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 001 (Experimental): TMC435 150 mg capsule once daily for 7 days (Trt A C D)
  Interventions: Drug: TMC435
- 002 (Experimental): erythromycin 500 mg tablets three times a day for 6 days + 1 morning dose for 7th day (Trt B)
  Interventions: Drug: erythromycin
- 003 (Experimental): erythromycin 500 mg tablets three times a day for 7 days (Trt C)
  Interventions: Drug: erythromycin
- 004 (Experimental): TMC435 50 mg capsule once daily for 7 days (Trt F)
  Interventions: Drug: TMC435
- 005 (Experimental): Darunavir 2 x 400 mg tablet once daily for 7 days (Trt E F)
  Interventions: Drug: Darunavir
- 006 (Experimental): Ritonavir 100 mg tablet once daily for 7 days (Trt E F)
  Interventions: Drug: Ritonavir

INTERVENTIONS:
Drug: erythromycin — 500 mg tablets three times a day for 6 days + 1 morning dose for 7th day (Trt B)
  Arms: 002
Drug: Ritonavir — 100 mg tablet once daily for 7 days (Trt E, F)
  Arms: 006
Drug: TMC435 — 150 mg capsule once daily for 7 days (Trt A, C, D)
  Arms: 001
Drug: Darunavir — 2 x 400 mg tablet once daily for 7 days (Trt E, F)
  Arms: 005
Drug: TMC435 — 50 mg capsule once daily for 7 days (Trt F)
  Arms: 004
Drug: erythromycin — 500 mg tablets three times a day for 7 days (Trt C)
  Arms: 003

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of erythromycin or DRV/r on the steady-state pharmacokinetics of TMC435, the effect of a steady-state concentration of TMC435 (150 mg) on the steady-state pharmacokinetics of erythromycin and the effect of a steady-state concentration of TMC435 (50 mg) on the steady-state pharmacokinetics of DRV/r. We will also study the short-term safety and tolerability of TMC435 given alone and given togehter with erythromycin (Panel 1) or DRV/r (Panel 2). Steady state is a term that means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body, and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for treatment of chronic hepatitis C virus (HCV) infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). Erythromycin is an antibiotic and Darunavir/ritonavir (DRV/r) is currently indicated for the treatment of HIV infection. TMC435 is metabolized by the degradation enzyme CYP3A. Erythromycin and DRV/r are respectively moderate and strong inhibitors of the degradation enzyme CYP3A. The result of this study will provide dosing recommendations for TMC435 and for erythromycin or DRV/r, when being coadministered. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (sequence of treatment with study medications is assigned by chance), crossover trial in 48 healthy volunteers to investigate the pharmacokinetic interaction between TMC435, at steady state, and DRV/r or erythromycin, at steady-state. The volunteers will be allocated to one of two panels. In Panel 1, volunteers will receive three treatments (Trts A, B and C) in a randomized order. Volunteers will receive TMC435 150 mg once daily for 7 days (Trt A) and erythromycin 500 mg three times daily for 6 days + a morning dose on day 7 (Trt B) and TMC435 150 mg once daily for 7 days + erythromycin 500 mg three tmes daily for 7 days (Trt C). In Panel 2, volunteers will receive three treatments (Trts D, E and F) in a randomized order. Volunteers will receive TMC435 150 mg once daily for 7 days (Trt D), DRV/r 800/100 mg once daily for 7 days (Trt E) and TMC435 50 mg once daily for 7 days + DRV/r 800/100 mg once daly for 7 days (Trt F). In both panels, there will be a washout period (a period when no study drug will be taken, in order to have all the medication eliminated from the body before starting a new treatment) of at least 10 (Panel 1) or 7 (Panel 2) days between last intake of the study medication in one session and the first intake of study medication in the subsequent session. Pharmacokinetic profiles of all four compounds (TMC435, DRV, ritonavir and erythromycin) will be determined through blood samples taken at regular intervals during the study. Safety and tolerability will be assessed during the study period and during follow up. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, on Day 1, Day 7 and Day 8 and at the follow up visit at 1 week after last dose of study medication in the last session. A physical examination will be performed at screening, on Day -1 (= day before first medication intake in each session for both panels) or Day 1, on Day 8 and during the follow-up visit. Volnteers will be admitted to the unit on Day-1, discharged on Day2, re-admitted on Day6 and discharged again on Day8. Each volunteer follows 3 treatment (Trt) periods, which are a minimum 10 days (Panel 1) or 7 days (Panel 2) apart from each other. All treatment periods take 7 days and all drugs are for oral intake. Panel 1: Trt A = 150 mg TMC435 once daily; Trt B = 500 mg erythromycin three times daily; Trt C: combining Trt A + B. Panel 2: Trt D = Trt A; Trt E = 800/100 mg DRV/r once daily; Trt D = 50 mg TMC435 once daily + Trt E.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests, vital signs, and electrocardiogram

Exclusion Criteria:

* Infection with hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* History of or any current medical condition which could impact the safety of the participant in the study
* Having previously been dosed with TMC435 in a multiple-dose trial with TMC435
* Having previously been dosed with TMC435 in more than 3 single-dose trials with TMC435

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-03; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in the steady-state plasma pharmacokinetics of TMC435 following co-administration with erythromycin (Panel 1). | Measured on Day 1 and Day 5-10 (Trt C). Reference for TMC435 is on Day 1 and Day 5-10 of Trt A.
Change in the steady-state plasma pharmacokinetics of TMC435 following co-administration with DRV/r (Panel 2). | Measured on Day 1 and Day 5-10 (Trt F). Reference for TMC435 is on Day 1 and Day 5-10 of Trt D.

SECONDARY OUTCOMES:
Change in the steady-state plasma pharmacokinetics of erythromycin following co-administration with TMC435 (Panel 1). | Measured on Day 1 and Day 5-7 (Trt C). Reference for erythromycin is on Day 1 and Day 5-7 of Trt B.
Change in the steady-state plasma pharmacokinetics of DRV/r following co-administration with TMC435 (Panel 2). | Measured on Day 1 and Day 5-8 (Trt F). Reference for DRV/r is on Day 1 and Day 5-8 of Trt E.
Number of participants with adverse events as a measure of safety and tolerability - TMC435 and erythromycin | Up to Day 67
Number of participants with adverse events as a measure of safety and tolerability - TMC435 and DRV/r | Up to Day 61

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Antwerp, Belgium